CLINICAL TRIAL: NCT00002704
Title: TREATMENT OF ISOLATED CNS RELAPSE OF ACUTE LYMPHOBLASTIC LEUKEMIA -- A PEDIATRIC ONCOLOGY GROUP-WIDE PHASE II STUDY
Brief Title: Radiation Therapy and Chemotherapy in Treating Children With CNS Relapse From Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01528; POG-9412; CDR0000064509 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-07-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2007-11

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia; TdT positive childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Filgrastim; Asparaginase; Cyclophosphamide; Daunorubicin; Dexamethasone; Etoposide; Leucovorin; Mercaptopurine; Mesna; Methotrexate; Hydrocortisone; Thiotepa; Vincristine

ARMS (1):
- Arm I (Experimental): Single Agent Chemotherapy. TSPA or DTC101. 3-Drug Combination Chemotherapy plus Triple Intrathecal Therapy. DM/DNR/VCR; plus TIT. 2-Drug Combination Chemotherapy plus Triple Intrathecal Therapy. ARA-C/ASP; plus TIT. 4-Drug Combination Chemotherapy with Leucovorin Rescue plus Triple Intrathecal Therapy. CTX/MP/MTX/VP-16; with CF; plus TIT. 3-Drug Combination Chemotherapy plus Triple Intrathecal Therapy. DM/DNR/VCR; plus TIT. 6-Drug Combination Chemotherapy with Leucovorin Rescue plus Triple Intrathecal Therapy. ARA-C/ASP/CTX/MP/MTX/VP-16; with CF; plus TIT. Radiotherapy plus 3-Drug Combination Chemotherapy. Craniospinal irradiation using x-rays with energies of 4-6 MV (electrons acceptable for spinal cord irradiation); plus ASP/DM/VCR. 2-Drug Combination Chemotherapy Alternating with 2-Drug Combination Chemotherapy. MP/MTX; alternating with CTX/VCR.
  Interventions: Biological: filgrastim; Drug: asparaginase; Drug: cyclophosphamide; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: etoposide; Drug: leucovorin calcium; Drug: liposomal cytarabine; Drug: mercaptopurine; Drug: mesna; Drug: methotrexate; Drug: therapeutic hydrocortisone; Drug: thiotepa; Drug: vincristine sulfate; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy

INTERVENTIONS:
Biological: filgrastim
Drug: asparaginase
Drug: cyclophosphamide
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: etoposide
Drug: leucovorin calcium
Drug: liposomal cytarabine
Drug: mercaptopurine
Drug: mesna
Drug: methotrexate
Drug: therapeutic hydrocortisone
Drug: thiotepa
Drug: vincristine sulfate
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
Phase II trial to study the effectiveness of radiation therapy following chemotherapy in treating children with CNS relapse from acute lymphoblastic leukemia. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with radiation therapy may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the efficacy and toxicity of intensified systemic treatment with delayed central nervous system (CNS) irradiation in children with acute lymphoblastic leukemia and isolated CNS disease.

II. Determine the efficacy of systemic thiotepa in reducing or clearing blasts in the cerebrospinal fluid of these patients.

III. Evaluate the toxicity of single dose thiotepa followed by dexamethasone, vincristine, daunorubicin, and triple intrathecal therapy in these patients.

IV. Determine the response rate of intrathecal sustained release cytarabine (DTC101) in patients with first bone marrow remission with first isolated CNS relapse.

V. Assess the safety and toxicity of DTC101 in these patients.

OUTLINE:

Patients with significant neurologic symptoms (e.g., seizures, cranial nerve palsy, paresis, mental status changes) are entered directly on the Induction regimen and do not receive the Therapeutic Window. The following acronyms are used: ARA-C Cytarabine, NSC-63878 ASP Asparaginase, NSC-109229 (E. coli) or 106977 (Erwinia) CF Leucovorin calcium, NSC-3590 CTX Cyclophosphamide, NSC-26271 DM Dexamethasone, NSC-34521 DNR Daunorubicin, NSC-82151 DTC101 Sustained release cytarabine G-CSF Granulocyte Colony-Stimulating Factor (Amgen), NSC-614629 HC Hydrocortisone, NSC-10483 Mesna Mercaptoethane sulfonate, NSC-113891 MP Mercaptopurine, NSC-755 MTX Methotrexate, NSC-740 TIT Triple Intrathecal Therapy, IT MTX/IT HC/IT ARA-C TMP-SMX Trimethoprim-sulfamethoxazole TSPA Thiotepa, NSC-6396 VCR Vincristine, NSC-67574 VP-16 Etoposide, NSC-141540

THERAPEUTIC WINDOW: Single Agent Chemotherapy. TSPA or DTC101. ** Thiotepa window closed as of 7/6/98 ** ** DTC101 window opened 11/15/99 **

INDUCTION: 3-Drug Combination Chemotherapy plus Triple Intrathecal Therapy. DM/DNR/VCR; plus TIT.

CONSOLIDATION: 2-Drug Combination Chemotherapy plus Triple Intrathecal Therapy. ARA-C/ASP; plus TIT.

INTENSIFICATION I: 4-Drug Combination Chemotherapy with Leucovorin Rescue plus Triple Intrathecal Therapy. CTX/MP/MTX/VP-16; with CF; plus TIT.

RE-INDUCTION: 3-Drug Combination Chemotherapy plus Triple Intrathecal Therapy. DM/DNR/VCR; plus TIT.

INTENSIFICATION II: 6-Drug Combination Chemotherapy with Leucovorin Rescue plus Triple Intrathecal Therapy. ARA-C/ASP/CTX/MP/MTX/VP-16; with CF; plus TIT.

CHEMORADIOTHERAPY: Radiotherapy plus 3-Drug Combination Chemotherapy. Craniospinal irradiation using x-rays with energies of 4-6 MV (electrons acceptable for spinal cord irradiation); plus ASP/DM/VCR.

MAINTENANCE: 2-Drug Combination Chemotherapy Alternating with 2-Drug Combination Chemotherapy. MP/MTX; alternating with CTX/VCR.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Acute lymphoblastic leukemia in first bone marrow remission (M1) with first isolated initial CNS relapse
* More than 5 WBC/microliter in cerebrospinal fluid (CSF) with blasts on cytospin OR immunophenotypic proof (encouraged) of relapse in CSF
* Identifiable blasts and presence on 2 CSF samples 3 weeks apart
* If B-cell terminal deoxynucleotidyl transferase (TdT) OR CD-10
* If T-cell TdT alone OR with CD-7

PATIENT CHARACTERISTICS:

* Age: Over 6 months and under 21 years at relapse
* Patients receiving sustained release cytarabine
* Performance status: Older than 10 years
* Karnofsky greater than 50% Less than 10 years
* Lansky greater than 50%
* Platelet count greater than 40,000/mm3
* Bilirubin less than 2.0 mg/dL
* SGPT less than 5 times normal
* Creatinine less than 1.5 times normal for age
* Normal metabolic parameters (serum electrolytes, calcium, and phosphorus)
* No clinical evidence of obstructive hydrocephalus, compartmentalization of the CSF flow, ventriculoperitoneal or ventriculoatrial shunt

PRIOR CONCURRENT THERAPY:

* Prior cumulative anthracycline dose less than 375 mg/sqm
* Patients receiving sustained release cytarabine
* At least 7 days since prior investigational drug
* At least 3 weeks since prior CNS directed therapy (6 weeks is prior nitrosourea)
* At least 1 week since intrathecal chemotherapy
* At least 8 weeks since prior craniospinal radiotherapy

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 1996-01; Primary Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio C. Barredo, MD, Study Chair — Medical University of South Carolina
Locations (70):
- United States (62):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - University of California Davis Medical Center, Sacramento, California
  - Children's Hospital and Health Center, San Diego, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - CCOP - Florida Pediatric, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Memorial Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Oklahoma Memorial Hospital, Oklahoma City, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - MBCCOP - South Texas Pediatric, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - McMaster Division, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico
- Switzerland (2):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Clinique de Pediatrie, Geneva

REFERENCES:
- [Background] Eapen M, Zhang MJ, Devidas M, Raetz E, Barredo JC, Ritchey AK, Godder K, Grupp S, Lewis VA, Malloy K, Carroll WL, Davies SM, Camitta BM; Children's Oncology Group; Center for International Blood and Marrow Transplant Research. Outcomes after HLA-matched sibling transplantation or chemotherapy in children with acute lymphoblastic leukemia in a second remission after an isolated central nervous system relapse: a collaborative study of the Children's Oncology Group and the Center for International Blood and Marrow Transplant Research. Leukemia. 2008 Feb;22(2):281-6. doi: 10.1038/sj.leu.2405037. Epub 2007 Nov 22. PMID 18033318
- [Result] Barredo JC, Devidas M, Lauer SJ, Billett A, Marymont M, Pullen J, Camitta B, Winick N, Carroll W, Ritchey AK. Isolated CNS relapse of acute lymphoblastic leukemia treated with intensive systemic chemotherapy and delayed CNS radiation: a pediatric oncology group study. J Clin Oncol. 2006 Jul 1;24(19):3142-9. doi: 10.1200/JCO.2005.03.3373. PMID 16809737